CLINICAL TRIAL: NCT02439021
Title: Effectiveness of the New Perilaryngeal Airway (CobraPLA™) in Comparison With the Laryngeal Mask Airway (LMA™) to Improve Oropharyngeal Leak Pressure Among Obese and Overweight Patients
Brief Title: Effectiveness of the New Perilaryngeal Airway in Comparison With the Laryngeal Mask Airway
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Assistant Professor, Department of Public Health, Qazvin University of Medical Sciences, Qazvin, Iran., Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 653
Record Dates: First submitted 2015-02-05; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- CobraPLA (Experimental): Patients will randomly assign to either LMA or Cobra PLATM
  Interventions: Device: COBRA
- LMA (Experimental): Patients will randomly assign to either LMA or Cobra PLATM
  Interventions: Device: LMA

INTERVENTIONS:
Device: COBRA
  Arms: CobraPLA
Device: LMA
  Arms: LMA

SUMMARY:
The Laryngeal Mask Airway (LMA) has been used widely for different patients and found to be highly safe for adult and pediatric patients. However, the LMA has some limitations and weaknesses (e.g. more insertion attempts in 5% to 10 % of all cases. Despite the easy insertion of the LMA, it is crucial to check correct placement of the LMA airway.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 to 35 kg/m2
* scheduled for surgery
* being older than 18 years
* Mallampati class I-III and BMI between 25 and 35

Exclusion Criteria:

* pregnancy
* morbid obese (BMI>35 kg/m2)
* a known difficult airway
* gastro-oesophageal reflux
* pharyngeal pathology
* emergency operation with full stomach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak | Up to 1 hours
Time to intubation | Up to 1 hours
  Time to intubation was measured from inserting of the device to the patient's month while connecting the breathing circuit

SECONDARY OUTCOMES:
successful intubation attempt | Up to 1 hours
  A successful intubation attempt was recognized if: the breathing circuit connected, the EtCO2 trace was revealed, and no air leak was detected at airway pressures of 15 cm H2O
incidence of sore throat | Up to 1 hours
incidence of dysphasia | Up to 1 hours
incidence of postoperative blood staining on mask | Up to 1 hours

CONTACTS AND LOCATIONS:
Overall Officials: Amir H Pakpour, PhD, Principal Investigator — Qazvin University Of Medical Sciences